CLINICAL TRIAL: NCT06859996
Title: A Comparison of Two Interventions for Chronic Cognitive Difficulties After mTBI
Brief Title: CORE (Cognitive Optimization Through Rehabilitation and Education) Study
Acronym: CORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Pagulayan, Associate Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00022262; 90DPHF0015-01-00 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Mild Traumatic Brain Injury; Concussion
Keywords: cognitive training; self-management; Veterans; concussion; psychoeducation; clinical trial
MeSH Terms: conditions — Brain Concussion | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- On-TRACC (Experimental)
  Interventions: Behavioral: Tools for Rehabilitation and Cognitive Care (On-TRACC)
- Brain Health Psychoeducation (Active Comparator)
  Interventions: Behavioral: Brain Health psychoeducation

INTERVENTIONS:
Behavioral: Tools for Rehabilitation and Cognitive Care (On-TRACC) — The On-TRACC intervention is administered one-on-one with a skilled clinician via telehealth and consists of an introductory session followed by 5 treatment sessions. Participants in the On-TRACC intervention will review various health and lifestyle factors that can affect cognitive functioning, learn and practice skills for managing cognitive and emotional symptoms, and develop personalized goals to support optimal cognitive functioning.
  Arms: On-TRACC
Behavioral: Brain Health psychoeducation — The Brain Health intervention is administered one-on-one with a skilled clinician via telehealth and consists of an introductory session followed by 5 treatment sessions. Participants in the Brain Health psychoeducation treatment will learn about various health and lifestyle factors that can affect brain health and cognitive functioning. In addition, they will be provided with resources and strategies for managing relevant factors and supporting optimal cognitive functioning.
  Arms: Brain Health Psychoeducation

SUMMARY:
Mild traumatic brain injury (mTBI) affects millions of individuals worldwide every year. It has long been thought that the vast majority of individuals who sustain a mTBI experience natural recovery with little or no intervention and return to baseline functioning within days to weeks of injury. However, recent large studies have demonstrated that a substantial number of individuals experience prolonged symptoms (e.g., cognitive impairment, headaches, affective symptoms). These symptoms, termed "Persistent Post-concussive Symptoms" (PPCS) are associated with significant functional disability and reduced quality of life (QOL) and can last for years post-injury. While PPCS can include affective, cognitive, and somatosensory/vestibular symptoms, objective and subjective cognitive symptoms - particularly in the domains of attention, memory, processing speed, and executive function - are among the most commonly reported following mTBI. There is currently no gold-standard intervention to address these symptoms. To address this gap, our research group developed a brief cognitive rehabilitation intervention called Tools for Rehabilitation and Cognitive Care (or On-TRACC).

The goals of this clinical trial are:

AIM 1: Compare the efficacy of On-TRACC to a psychoeducation control on reduction of self-reported cognitive post-concussive symptoms (Aim 1.1) and overall neurobehavioral post concussive symptoms and (Aim 1.2) following treatment and at 3-month follow-up (Aim 1.3) in a randomized clinical trial of community-dwelling adults with mTBI.

AIM 2: Compare the efficacy of On-TRACC and psychoeducation on change in secondary outcomes, including cognitive self-efficacy, compensatory strategy use, self-management skills, and quality of life at post-treatment and 3-month follow-up.

Exploratory AIM 3: Compare the efficacy of On-TRACC and psychoeducation on: primary and secondary outcomes at 6-months post-treatment and (Aim 3.1) explore whether engaging in On-TRACC leads to subsequent engagement in care by assessing whether there is a different level of participation in optional intervention booster sessions in the post-intervention period (Aim 3.2).

All participants will:

* Complete a series of assessments
* Complete 6 treatment sessions via telehealth (either On-TRACC or psychoeducation)

All participants will have the option of:

* Attending weekly "Booster Sessions" between 3 and 6-months post-treatment
* Completing neuropsychological assessments at 2 timepoints during the study

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Evidence of self-reported mTBI sustained in adulthood at least 3 months prior to the date of study enrollment (clinical discretion allowed for mTBI in late adolescence) AND documentation of diagnosed or suspected mTBI as defined by American Congress of Rehabilitation Medicine (ACRM) criteria in the medical record (e.g., on the problem list, has a diagnosis, encounter for a TBI, diagnosis via a TBI evaluation, or documented in a clinical note, etc).
* Endorsement of at least moderate symptoms (score of 3 or higher) on at least one of the cognitive items (forgetfulness, poor concentration, taking longer to think) from the Rivermead Postconcussion Symptom Questionnaire.
* Ability to read, speak and understand English enough to participate in healthcare in English without a translator.
* Willingness to participate in audio-recorded treatment sessions.
* Willingness to be randomized to treatment condition.
* Willingness to use clinical video teleconferencing (CVT) for research appointments (including be on camera for treatment sessions).
* Able to use and have access to a smart phone, tablet, or computer with internet access in private setting for treatment sessions.

Exclusion Criteria:

* History of neurologic injury or illness other than mTBI that can affect cognitive functioning (e.g., any lifetime severe TBI [Glasgow Coma Score (GCS)<=8; loss of consciousness (LOC)> 1 hour; posttraumatic amnesia (PTA)>1 week], seizure disorder, multiple sclerosis, neurodegenerative disorder).
* Alcohol abuse (operationalized as scoring 15 or more if male or 13 or more if female on the Alcohol Use Disorders Identification Test), or high-risk illicit drug use (as defined by modified Tobacco, Alcohol, Prescription Medications and Substance Use/Misuse (TAPS) Tool subscale scores > 2) in the past 3 months. Indication of alcohol/drug abuse or dependence in medical record is also sufficient to meet this exclusion criteria, per PI discretion.
* Active suicidal ideation/intent indicating significant risk, per PI discretion.
* Unstable medical or psychiatric condition (e.g., mania, psychotic symptoms) that would interfere with study participation.
* Behavioral issues noted in the record or observed during the screening process that would interfere with appropriate or safe CVT participation or study procedures.
* Prior participation in the On-TRACC intervention.
* Significant cognitive impairment that would limit ability to engage in treatment (as indicated by more than 1 error on a 6-item screener).
* Planned life events that would interfere with study participation during active treatment phase (e.g., major surgery, moving out of state, extended travel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory Total Score | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Measure of post-concussive symptoms
Neurobehavioral Symptom Inventory Cognitive Subscale Score | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Cognitive post-concussive symptoms

SECONDARY OUTCOMES:
Cognitive Concerns Self-Efficacy Scale | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Measure of perceived ability to effectively manage cognitive concerns and their impact on daily life
Compensatory Cognitive Strategies Scale | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Measure of frequency of compensatory strategy use
Patient Global Impression of Change | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Measure of symptoms and overall quality of life
Quality of Life After Brain Injury | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Measure of health-related quality of life after brain injury
Self-Management Assessment Scale | Pre-treatment, Immediately post-treatment, 3-months post-treatment
  Measure of ability to self-manage health

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pagulayan, PhD, Principal Investigator — University of Washington; Rhonda Williams, PhD, Principal Investigator — VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will submit all deidentified data from this study to the Inter-university Consortium for Political and Social Research (ICPSR) data repository for other researchers to use in future studies.
URL: https://www.icpsr.umich.edu/web/pages/

REFERENCES:
- [Background] Pagulayan KF, Rau HK, Sheppard DP, Shulein OM, Onstad-Hawes E, Hoffman JM, Williams RM. On-TRACC Pilot Study: A Novel Intervention for Persistent Post-Concussive Cognitive Symptoms. J Head Trauma Rehabil. 2025 Jul-Aug 01;40(4):E308-E319. doi: 10.1097/HTR.0000000000001014. Epub 2024 Sep 29. PMID 39853212
- See also: Dr. Pagulayan's Research Website — https://sites.uw.edu/farkat/